CLINICAL TRIAL: NCT00487227
Title: Levels of Caffeine Lower Than Those Found in Decaffeinated Beverages Exert Effects on Cognition, Mood, and Autonomic Activity
Brief Title: Effects of Low Doses of Caffeine on Mood, Physiology and Mental Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 7G2CDCH
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: caffeine; coffee; decaffeinated; cognition; mood; autonomic
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 2.5mg caffeine (Experimental)
  Interventions: Drug: caffeine
- 5mg caffeine (Experimental)
  Interventions: Drug: caffeine
- 10mg caffeine (Experimental)
  Interventions: Drug: caffeine

INTERVENTIONS:
Drug: caffeine
  Arms: 10mg caffeine; 2.5mg caffeine; 5mg caffeine
Drug: Placebo
  Arms: Placebo

SUMMARY:
It is often assumed that levels of caffeine found in 'decaffeinated' beverages are below any psychopharmacological threshold. However, recent findings indicate that caffeine doses as low as 9 mg may be psychoactive. The effects of caffeine have also been shown up to 6 hours post-administration. The study aimed to establish the lowest active dose of caffeine, and to ascertain the duration of any effects.

DETAILED DESCRIPTION:
The majority of recent caffeine studies have evaluated doses in the range of 75 - 150 mg or 1 - 2 mg/kg (approximately 130 - 260 ml fresh coffee). Such doses produce well characterised effects; including increased 'alertness', and improvements to measures of reaction time and sustained attention. A previous study has demonstrated improvements to performance following 9 mg caffeine, which represents the lowest known psychoactive dose of caffeine. A number of these effects, including elevated salivary caffeine levels, were still apparent at 6 hours post-caffeine consumption (9). Findings showing effects of 12.5 and 9 mg caffeine are important as these are approaching the levels found in decaffeinated beverages, which are assumed to have no behavioural or physiological effects. However, despite extensive research in this area, the lower threshold for psychoactive effects has not been established. A randomised, placebo-controlled, double-blind, balanced crossover study was undertaken. 20 young men and women (13 female, mean age 20.7 years, standard deviation 2.4) undertook computerised assessments of memory and attention and rated subjective mood. Autonomic activity and salivary caffeine were co-monitored. Assessment took place at baseline, 1, 3, 6, and 9 hours post-administration of placebo, 2.5, 5, and 10 mg caffeine (on separate days) administered in 150 ml fruit juice.

ELIGIBILITY:
Inclusion Criteria:

* native English speaker

Exclusion Criteria:

* pregnancy
* medication
* anaemia
* heart disorder
* diabetes
* respiratory disorder
* epilepsy
* asthma
* panic attacks
* habitual smoking
* food allergy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-06; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline speed of attention | 1 hour
Change from baseline speed of attention | 3 hours
Change from baseline speed of attention | 6 hours
Change from baseline speed of attention | 9 hours

SECONDARY OUTCOMES:
Change from baseline accuracy of attention | 1 hour
Change from baseline accuracy of attention | 3 hours
Change from baseline accuracy of attention | 6 hours
Change from baseline accuracy of attention | 9 hours
Change from baseline speed of memory | 1 hour
Change from baseline speed of memory | 3 hours
Change from baseline accuracy of memory | 6 hours
Change from baseline accuracy of memory | 9 hours
Change from baseline subjective mood | 1 hour
Change from baseline subjective mood | 3 hours
Change from baseline subjective mood | 6 hours
Change from baseline subjective mood | 9 hours
Change from baseline blood pressure | 1 hour
Change from baseline blood pressure | 3 hours
Change from baseline blood pressure | 6 hours
Change from baseline blood pressure | 9 hours
Change from baseline heart rate | 1 hour
Change from baseline heart rate | 3 hours
Change from baseline heart rate | 6 hours
Change from baseline heart rate | 9 hours
Change from baseline salivary caffeine levels | 1 hour
Change from baseline salivary caffeine levels | 3 hours
Change from baseline salivary caffeine levels | 6 hours
Change from baseline salivary caffeine levels | 9 hours

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Scholey, Principal Investigator — Northumbria University